CLINICAL TRIAL: NCT07214844
Title: A Prospective, Randomized, Assessor Blind, Active-controlled, Single-center Study to Evaluate the Efficacy of Iovera Lumbar Medial Branch Cryoneurolysis Versus Radiofrequency Ablation for the Treatment of Facet-mediated Chronic Low Back Pain
Brief Title: A Prospective Study to Evaluate the Efficacy of Iovera Lumbar Medial Branch Cryoneurolysis Versus Radiofrequency Ablation for the Treatment of Chronic Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-16365; CRS-133 (Other: Pacira Pharmaceuticals Inc.)
Record Dates: First submitted 2025-10-06; First posted 2025-10-09 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Low Back Pain, Chronic
Keywords: Iovera; Radiofrequency ablation; cryoneurolysis; low back pain; lumbar medial branch
MeSH Terms: conditions — Low Back Pain; Bronchiolitis Obliterans Syndrome | interventions — Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- iovera cryoneurolysis (Experimental): Subjects will receive iovera cryoneurolysis to the medial branch nerves of the lumbar spine.
  Interventions: Device: Iovera Medial Branch Cryoneurolysis
- Radiofrequency ablation (RFA) (Active Comparator): Subjects will receive radiofrequency ablation (RFA) to the medial branch nerves of the lumbar spine.
  Interventions: Procedure: Radiofrequency ablation (RFA)

INTERVENTIONS:
Device: Iovera Medial Branch Cryoneurolysis — The iovera group will receive fluoroscopic guided medial branch cryoneurolysis with the subject in the prone position under asepsis:
  * Investigator injects 1% lidocaine at the treatment site using a 25-gauge, 3/4 -inch needle to numb the skin and tissue around the facet joint
  * Introducer needle is inserted through the skin wheal to the target medial branch nerve below the junction of the superior articular and transverse process
  * The introducer needle is positioned, and an x-ray image is taken to confirm the needle's position
  * With the desired introducer needle position confirmed, the iovera Smart Tip is guided through the introducer needle and the handpiece is secured to the Smart Tip. The start/stop button on the iovera° handpiece is then pressed to start the cycle.
  * After the cycle is complete, Smart Tip can be removed and next treatment cycle can commence ensuring an overlap of the ice ball
  * The needle is removed, and light compression is applied with gauze
  Arms: iovera cryoneurolysis
Procedure: Radiofrequency ablation (RFA) — Subjects will receive a fluoroscopic guided RFA medial branch block in the prone position under asepsis:
  * The Right L4, L5, S1 articular pillars are identified with fluoroscopy at each level and the target points are located
  * A skin wheal is formed using 5mL 1% Lidocaine and 5mL 0.25% Bupivacaine
  * A 20-gauge, 10cm needle with a 10mm active tip is inserted using a 15-degree oblique view and a 15-degree caudad angle onto the waist of each pillar at each level
  * Anterior-posterior and oblique neuroforamen views confirm positioning
  * Stimulation is performed and recorded to confirm proper needle placement
  * A mixture of 3mL of 0.25% Bupivacaine and 2mL of 1% Lidocaine is divided and injected at each level
  * A lesion is then performed at each level at 80 degrees centigrade for 60 seconds
  * The needles are removed, and bandages applied to the puncture sites
  * The same procedure is carried out on the opposite side
  Arms: Radiofrequency ablation (RFA)

SUMMARY:
A research study is being conducted to compare two treatments for long-term low back pain:

* One uses the iovera° system, which applies cold to certain nerves in the lower back.
* The other is the standard treatment called radiofrequency ablation, which uses heat.

The primary objective is to find out which treatment works better to reduce back pain. Participants in this study will be randomly placed in one of the two treatment groups. The clinical research team will check on participant pain levels and overall health before and after the procedure for about 12 months. The entire study will last about 14 months for each participant.

DETAILED DESCRIPTION:
Secondary objectives of this study include:

1. Evaluate safety outcomes (i.e., adverse device effects, serious adverse device effects, and adverse events) related to iovera° treatment;
2. Evaluate clinical outcomes related to iovera° treatment including pain, functional disability, and concomitant medication use (including opioids and analgesics);
3. Evaluate the treatment success and failure rate of iovera° medial branch cryoneurolysis;
4. Evaluate health-related quality of life (HRQoL);
5. Evaluate subject satisfaction with pain management;
6. Identify subgroups of patients who are most and least likely to benefit from iovera° medial branch cryoneurolysis for facet-mediated CLBP.

An adaptive study design will be used in this study. A blinded interim analysis will occur after approximately 56 total subjects, at least 28 per study arm, have completed assessment data for the primary efficacy outcome. The primary purpose of this interim analysis is to evaluate the sample size assumptions.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for participation:

* Subjects at least 18 years of age at Screening
* Primary complaint of axial low-back pain suggestive of bilateral facet joint involvement (i.e., facet mediated CLBP) by evidence of provocative testing (e.g., axial loading, paraspinal tenderness)
* Low back pain is chronic (i.e., ≥ 3 months' duration)
* Low back pain is moderate to severe (score of ≥ 5 to ≤ 9) on the 0 to 10 NRS at Screening
* Low back pain causes functional impairment (≥ 30% on ODI) at Screening
* Successful trial of two diagnostic medial branch blocks consisting of two positive blocks with local anesthetic only (i.e., no steroids) that results in at least 80% relief of primary (index) pain for the duration of the local anesthetic used
* Failure of at least three months of conservative non-operative therapy (e.g., physical therapy, chiropractic care, sleep hygiene, weight loss, spinal injections, NSAIDs, physician-directed exercise program or other appropriate analgesics)
* Able to provide informed consent, adhere to the study visit schedule, and complete all study assessment

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria will not be eligible for participation in this study:

* Active workers' compensation, personal injury, Social Security disability insurance (SSDI), or other litigation/compensation related to the spine
* Serious spinal disorders (verified on magnetic resonance imaging (MRI)) that may impact outcomes, including any of the following:

  1. Suspected cauda equina syndrome (e.g., bowel/bladder dysfunction)
  2. Infection
  3. Tumor
  4. Traumatic fracture
  5. Systemic inflammatory spondyloarthropathy
  6. Lumbar radiculopathy/radiculitis (i.e., root irritation and deficit)
  7. Neurogenic claudication Prior lumbar spinal fusion surgery at the intended treatment levels
* Comorbidity that, in the judgment of the Investigator, may affect the subject's ability to participate in the study including lumbar radiculopathy and neuropathic pain disorder
* Currently pregnant, nursing, or planning to become pregnant during the study
* Known contraindication to study device, including any of the following:

  1. Cryoglobulinemia
  2. Paroxysmal cold hemoglobinuria
  3. Cold urticaria
  4. Raynaud's disease
  5. Open and/or infected wounds at or near the treatment site
  6. Coagulopathy
* Severe chronic pain disorder that in the opinion of the investigator may impact study outcomes
* Presence of any of the following:

  1. Spinal neurostimulator
  2. Intrathecal analgesic drug pump
  3. Cardiac implantable device
* Current manifestation of poorly controlled mental illness or catastrophizing that in the opinion of the investigator may meaningfully impact treatment outcomes, including any of the following:

  1. Mood disorder (e.g., depression, bipolar)

     Patient Health Questionnaire (PHQ-9) ≥ 12 at Screening
  2. Psychotic disorder (e.g., schizophrenia)
  3. Catastrophizing

Patient Catastrophizing Scale (PCS) score > 30 at Screening

* Subject received other spine intervention/therapies in the 30 days prior to block administration (e.g., spinal injections, minimally invasive therapies, surgical therapies) at the intended lumbar treatment levels
* Subject received radiofrequency ablation in the low back region ≤ 6 months before study enrollment at the intended lumbar treatment levels
* Pain relief following diagnostic medial branch blocks lasted longer than the duration of the local anesthetic used (i.e., > 24 hours)

  1. History, suspicion, or clinical manifestation of:
  2. Alcohol abuse or dependence
  3. Illicit drug use
* Opioid abuse or dependence (≥40 mg medication PO/day in past 30 days)
* Given the COVID-19 pandemic, the subject must be medically fit/cleared for surgery by the investigator. If there is a concern about a subject's recent or potential exposure to COVID-19, or if the subject is not medically fit/cleared for surgery due to suspected COVID-19 illness/symptoms (or other serious illness), the subject must be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Numeric rating scale (NRS) pain intensity score | 360 days after intervention
  Subjects will evaluate their pain in the low back region using an 11-point NRS where 0=no pain and 10=worst possible pain, such that higher scores are associated with greater pain intensity.
  * Pain intensity scores (using the NRS) measured as "On a scale from 0 to 10, where 0 equals no pain and 10 equals the worst possible pain, how much pain are you experiencing in your low back right now?
  * Pain intensity scores (using the numeric rating scale; NRS) measured as "On a scale from 0 to 10, where 0 equals no pain and 10 equals the worst possible pain, what was the worst pain in your low back in the last 24 hours?"
  * Pain intensity scores (using the NRS) measured as "On a scale from 0 to 10, where 0 equals no pain and 10 equals the worst possible pain, what was the average pain in your low back in the last 24 hours?"
  Mean numeric pain intensity rating scores will be summarized by study arm using basic descriptive statistics.

SECONDARY OUTCOMES:
Change in Functional Disability from baseline using Oswestry Disability Questionnaire | 360 days after intervention
  The Oswestry Disability Questionnaire is a 10-item condition-specific measure of functional status (pain and disability) for patients with low back pain (LBP). Each question has 6 possible answers (0 = worse, 5 = best). The raw score is doubled to provide a percent score from 0 to 100%; with 0 equaling no disability and 100% equaling the worst possible outcome. It measures pain-related disability. Change from baseline scores will be summarized by study arm using descriptive statistics.
Change in Patients' Global Impression of Change (PGIC) scale from baseline | 360 days after intervention
  The Patient Global Impression of Change (PGIC) scale is a subjective measure used to evaluate a patient's perceived improvement following treatment, rated on a 7-point Likert scale ranging from 1 to 7 [1= "No change (or condition has got worse)" to 7 = "a great deal better, and a considerable improvement that has made all the difference"], wherein higher scores are associated with improved patient impression following treatment. Change from baseline scores will be summarized by study arm using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Karina Gritsenko, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Multidisciplinary Pain Program, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wray JK, Dixon B, Przkora R. Radiofrequency Ablation. 2023 Jun 12. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK482387/ PMID 29494009
- [Background] Winston P, Mills PB, Reebye R, Vincent D. Cryoneurotomy as a Percutaneous Mini-invasive Therapy for the Treatment of the Spastic Limb: Case Presentation, Review of the Literature, and Proposed Approach for Use. Arch Rehabil Res Clin Transl. 2019 Oct 17;1(3-4):100030. doi: 10.1016/j.arrct.2019.100030. eCollection 2019 Dec. PMID 33543059
- [Background] Tetzlaff W, Bisby MA. Neurofilament elongation into regenerating facial nerve axons. Neuroscience. 1989;29(3):659-66. doi: 10.1016/0306-4522(89)90138-3. PMID 2500618
- [Background] Starr JB, Gold L, McCormick Z, Suri P, Friedly J. Trends in lumbar radiofrequency ablation utilization from 2007 to 2016. Spine J. 2019 Jun;19(6):1019-1028. doi: 10.1016/j.spinee.2019.01.001. Epub 2019 Jan 10. PMID 30639589
- [Background] Shaffer JP, Williams VB, Shin SS. Cryoneurolysis for Digital Neuralgia in Professional Baseball Players: A Case Series. Orthop J Sports Med. 2022 May 12;10(5):23259671221096095. doi: 10.1177/23259671221096095. eCollection 2022 May. PMID 35601731
- [Background] Sayed D, Grider J, Strand N, Hagedorn JM, Falowski S, Lam CM, Tieppo Francio V, Beall DP, Tomycz ND, Davanzo JR, Aiyer R, Lee DW, Kalia H, Sheen S, Malinowski MN, Verdolin M, Vodapally S, Carayannopoulos A, Jain S, Azeem N, Tolba R, Chang Chien GC, Ghosh P, Mazzola AJ, Amirdelfan K, Chakravarthy K, Petersen E, Schatman ME, Deer T. The American Society of Pain and Neuroscience (ASPN) Evidence-Based Clinical Guideline of Interventional Treatments for Low Back Pain. J Pain Res. 2022 Dec 6;15:3729-3832. doi: 10.2147/JPR.S386879. eCollection 2022. PMID 36510616
- [Background] Rubin DI. Epidemiology and risk factors for spine pain. Neurol Clin. 2007 May;25(2):353-71. doi: 10.1016/j.ncl.2007.01.004. PMID 17445733
- [Background] Rubenstein J, Harvey AW, Vincent D, Winston P. Cryoneurotomy to Reduce Spasticity and Improve Range of Motion in Spastic Flexed Elbow: A Visual Vignette. Am J Phys Med Rehabil. 2021 May 1;100(5):e65. doi: 10.1097/PHM.0000000000001624. No abstract available. PMID 33105153
- [Background] Radnovich R, Scott D, Patel AT, Olson R, Dasa V, Segal N, Lane NE, Shrock K, Naranjo J, Darr K, Surowitz R, Choo J, Valadie A, Harrell R, Wei N, Metyas S. Cryoneurolysis to treat the pain and symptoms of knee osteoarthritis: a multicenter, randomized, double-blind, sham-controlled trial. Osteoarthritis Cartilage. 2017 Aug;25(8):1247-1256. doi: 10.1016/j.joca.2017.03.006. Epub 2017 Mar 20. PMID 28336454
- [Background] Perolat R, Kastler A, Nicot B, Pellat JM, Tahon F, Attye A, Heck O, Boubagra K, Grand S, Krainik A. Facet joint syndrome: from diagnosis to interventional management. Insights Imaging. 2018 Oct;9(5):773-789. doi: 10.1007/s13244-018-0638-x. Epub 2018 Aug 8. PMID 30090998
- [Background] Mehta CR, Pocock SJ. Adaptive increase in sample size when interim results are promising: a practical guide with examples. Stat Med. 2011 Dec 10;30(28):3267-84. doi: 10.1002/sim.4102. Epub 2010 Nov 30. PMID 22105690
- [Background] Manchikanti L, Singh V, Datta S, Cohen SP, Hirsch JA; American Society of Interventional Pain Physicians. Comprehensive review of epidemiology, scope, and impact of spinal pain. Pain Physician. 2009 Jul-Aug;12(4):E35-70. PMID 19668291
- [Background] Manchikanti L, Kaye AD, Soin A, Albers SL, Beall D, Latchaw R, Sanapati MR, Shah S, Atluri S, Abd-Elsayed A, Abdi S, Aydin S, Bakshi S, Boswell MV, Buenaventura R, Cabaret J, Calodney AK, Candido KD, Christo PJ, Cintron L, Diwan S, Gharibo C, Grider J, Gupta M, Haney B, Harned ME, Helm Ii S, Jameson J, Jha S, Kaye AM, Knezevic NN, Kosanovic R, Manchikanti MV, Navani A, Racz G, Pampati V, Pasupuleti R, Philip C, Rajput K, Sehgal N, Sudarshan G, Vanaparthy R, Wargo BW, Hirsch JA. Comprehensive Evidence-Based Guidelines for Facet Joint Interventions in the Management of Chronic Spinal Pain: American Society of Interventional Pain Physicians (ASIPP) Guidelines Facet Joint Interventions 2020 Guidelines. Pain Physician. 2020 May;23(3S):S1-S127. PMID 32503359
- [Background] Katz JN. Lumbar disc disorders and low-back pain: socioeconomic factors and consequences. J Bone Joint Surg Am. 2006 Apr;88 Suppl 2:21-4. doi: 10.2106/JBJS.E.01273. PMID 16595438
- [Background] GBD 2017 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 354 diseases and injuries for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1789-1858. doi: 10.1016/S0140-6736(18)32279-7. Epub 2018 Nov 8. PMID 30496104
- [Background] Evans PJ, Lloyd JW, Green CJ. Cryoanalgesia: the response to alterations in freeze cycle and temperature. Br J Anaesth. 1981 Nov;53(11):1121-7. doi: 10.1093/bja/53.11.1121. PMID 7326160
- [Background] Dasa V, Lensing G, Parsons M, Harris J, Volaufova J, Bliss R. Percutaneous freezing of sensory nerves prior to total knee arthroplasty. Knee. 2016 Jun;23(3):523-8. doi: 10.1016/j.knee.2016.01.011. Epub 2016 Feb 10. PMID 26875052
- [Background] Cohen SP, Raja SN. Pathogenesis, diagnosis, and treatment of lumbar zygapophysial (facet) joint pain. Anesthesiology. 2007 Mar;106(3):591-614. doi: 10.1097/00000542-200703000-00024. PMID 17325518
- [Background] Cohen SP, Bhaskar A, Bhatia A, Buvanendran A, Deer T, Garg S, Hooten WM, Hurley RW, Kennedy DJ, McLean BC, Moon JY, Narouze S, Pangarkar S, Provenzano DA, Rauck R, Sitzman BT, Smuck M, van Zundert J, Vorenkamp K, Wallace MS, Zhao Z. Consensus practice guidelines on interventions for lumbar facet joint pain from a multispecialty, international working group. Reg Anesth Pain Med. 2020 Jun;45(6):424-467. doi: 10.1136/rapm-2019-101243. Epub 2020 Apr 3. PMID 32245841
- [Background] Chou R, Atlas SJ, Stanos SP, Rosenquist RW. Nonsurgical interventional therapies for low back pain: a review of the evidence for an American Pain Society clinical practice guideline. Spine (Phila Pa 1976). 2009 May 1;34(10):1078-93. doi: 10.1097/BRS.0b013e3181a103b1. PMID 19363456
- [Background] Cassidy JD, Carroll LJ, Cote P. The Saskatchewan health and back pain survey. The prevalence of low back pain and related disability in Saskatchewan adults. Spine (Phila Pa 1976). 1998 Sep 1;23(17):1860-6; discussion 1867. doi: 10.1097/00007632-199809010-00012. PMID 9762743
- [Background] Birkenmaier C, Veihelmann A, Trouillier H, Hausdorf J, Devens C, Wegener B, Jansson V, von Schulze Pellengahr C. Percutaneous cryodenervation of lumbar facet joints: a prospective clinical trial. Int Orthop. 2007 Aug;31(4):525-30. doi: 10.1007/s00264-006-0208-6. Epub 2006 Aug 23. PMID 16927087
- [Background] Barnard D. The effects of extreme cold on sensory nerves. Ann R Coll Surg Engl. 1980 May;62(3):180-7. PMID 7396346